CLINICAL TRIAL: NCT03428776
Title: Timeliness of Immunization and Compliance Assessment Study
Acronym: TICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Bal Umang Drishya Sanstha (BUDS), India (Other); Royal Datamatics Pvt. Ltd. (RDPL), India (Unknown); St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00161339
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Vaccinations

STUDY DESIGN:
Intervention Model Description: Single blinded prospective study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controls (Sham Comparator): Self returns
  Interventions: Other: Record keeping
- Standard Compliance-linked incentives (Active Comparator): Standard mobile-phone reminders and compliance-linked incentives
  Interventions: Behavioral: Standard Compliance-linked incentives
- Intelligent Compliance-linked incentives (Active Comparator): Intelligent mobile-phone reminders and compliance-linked incentives
  Interventions: Behavioral: Intelligent Compliance-linked incentives

INTERVENTIONS:
Behavioral: Standard Compliance-linked incentives — Standard mobile-phone reminders and compliance-linked incentives Electronic immunization records on cloud-based software platform and use of biometric identification
  Arms: Standard Compliance-linked incentives
Behavioral: Intelligent Compliance-linked incentives — Intelligent mobile-phone reminders and compliance-linked incentives Electronic immunization records on cloud-based software platform and use of biometric identification
  Arms: Intelligent Compliance-linked incentives
Other: Record keeping — Electronic immunization records on cloud-based software platform and use of biometric identification
  Arms: Controls

SUMMARY:
Although coverage for primary childhood immunizations has improved, a significant proportion of young children and pregnant women living in low-resource settings remain inadequately immunized. While young children receive some primary vaccines, many are never fully vaccinated. Progressive decline in immunizations are in large part attributable to poor follow-up and compliance. Major challenges include maintaining immunization records linked to positive identification of the individual child, incentivizing follow-up and return immunizations and efficiently identifying and targeting non-compliant subjects. Mobile-phone costs have decreased dramatically in the developing world with rapid proliferation of web and mobile-phone connectivity. Novel approaches that integrate these modern technologies with existing resources in low and middle income countries can cost-effectively address these challenges. In this proposal, investigators will evaluate a novel software platform, utilizing biometric identification and of subjects, paired with intelligent and subject-aware, mobile-phone reminders and compliance-linked incentives to improve uptake and coverage of primary vaccinations in young children.

DETAILED DESCRIPTION:
A cloud-based, biometric-linked vaccination record, mobile-phone reminder and compliance-linked incentive software platform to provide robust and universal access of vaccinations. The investigators will implement this platform in a low-resource settings with the following features: a) Cloud-based for robust and universal access. b) Biometric-linked for positive identification. c) Digital storage and reporting for transparent view of program operations. d) Global Positioning System (GPS)-linked, allowing rapid assessment of vaccination status of communities. e) Increasing vaccination uptake and coverage by intelligent and subject-aware automated reminders and compliance-linked incentives.

ELIGIBILITY:
Inclusion Criteria:

* Mother (or caregiver) with one or more children ≤24 months in their family will be enrolled
* There will be no exclusion criteria based on race, ethnicity or gender.

Exclusion Criteria:

- Participants unable or unwilling to comply with the protocol or with any other condition that would impede compliance or hinder completion of the study (e.g. no mobile-phone in the family), or failure to give informed consent would be the only exclusion criteria.

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2065 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Timeliness of immunization | 12-15 months
  Defined as the proportion of immunizations administered before the scheduled date or within 14 days of the after scheduled date.

SECONDARY OUTCOMES:
Immunization rate | 12-15 months
  Calculated for each individual child and defined as the proportion of the total number of immunizations received divided by the total number of immunizations required at the time of measurement (e.g. at enrollment, end of study, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Jain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- BUDS, Haryāna, India